CLINICAL TRIAL: NCT04014166
Title: Study of Human Umbilical Cord-derived Mesenchymal Stem Cells for Treatment of Refractory Immune Thrombocytopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC2019002
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-06

CONDITIONS: Thrombocytopenia; Mesenchymal Stem Cells
Keywords: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15 refractory ITP patients (Experimental): 15 enrolled refractory ITP patients will be picked up to infuse hUC-MSCs at the indicated dose.
  Interventions: Other: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)

INTERVENTIONS:
Other: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) — This is a single-arm study to evaluate the safety and efficacy of hUC-MSCs to treat refractory immune thrombocytopenia. The dose of hUC-MSCs will be successively divided into three increasing dose(group A: hUC-MSCs 0.5×10^6/kg, weekly for 4 weeks, 3 patients; group B: hUC-MSCs 1.0×10^6/kg, weekly for 4 weeks, 3 patients; hUC-MSCs 2.0×10^6/kg, weekly for 4 weeks, 3 patients) with 3 patients in each group according to the dose. The principle of increasing dose will be carried out successively from low dose to high dose group. According to the results of the safety and efficacy data from these 9 patients, the investigator will determine one of the doses and expand the sample size to 6 cases.

SUMMARY:
Primary Objective: To evaluate the safety and efficacy of human umbilical cord-derived mesenchymal stem cells（hUC-MSCs） to treat refractory immune thrombocytopenia（ITP）.

Secondary Objective: To observe the changes of immune function in refractory ITP patients with human umbilical cord-derived mesenchymal stem cells（hUC-MSCs） after infusion, and to explore and reveal the mechanism of hUC-MSCs in treating ITP.

DETAILED DESCRIPTION:
Human umbilical cord (hUC)-derived mesenchymal stem cells (MSCs) have been shown to have marked therapeutic effects in a number of inflammatory diseases and autoimmune diseases in humans based on their potential for immunosuppression and their low immunogenicity. Currently, no more data is available on the safety and effectiveness of hUC-MSCs to treat immune thrombocytopenia patients.

This is a single-arm study to evaluate the safety and efficacy of hUC-MSCs to treat refractory immune thrombocytopenia（ITP）. In addition, it is the objective of this study to observe the changes of immune function in refractory ITP patients after hUC-MSCs infusion, and to explore and reveal the mechanism of hUC-MSCs in treating ITP.

The investigator will assess the changes of the platelet counts after hUC-MSCs infusion from week 1 to week 28, and observe incidence of adverse events during and after hUC-MSCs infusion.The investigator will complete virus detection( including HBV, HCV, HIV, Syphilis, etc) at week 4 and week 16 after hUC-MSCs infusion.

The dose of hUC-MSCs will be successively divided into three increasing dose(group A: hUC-MSCs 0.5×10^6/kg, weekly for 4 weeks, 3 patients; group B: hUC-MSCs 1.0×10^6/kg, weekly for 4 weeks, 3 patients; hUC-MSCs 2.0×10^6/kg, weekly for 4 weeks, 3 patients) with 3 patients in each group according to the dose.

The principle of increasing dose will be carried out successively from low dose to high dose group. According to the results of the safety and efficacy data from these 9 patients, the investigator will determine one of the doses and expand the sample size to 6 cases.

The investigator will observe the concentration of hUC-MSCs in peripheral blood from female patients after the first hUC-MSCs infusion at 10 time points, including 30 minutes before hUC-MSCs infusion, 30 minutes, 60 minutes, 2 hours, 4 hours, 8 hours, 16 hours, 24 hours,48 hours and 96 hours after the first hUC-MSCs infusion.

The investigator will detect antibody production of hUC-MSCs in peripheral blood from the first 9 patients at 2 time points, including 30 minutes before the first hUC-MSCs infusion and 48 hours after the last hUC-MSCs infusion.

The investigator will observe the changes of immune function in refractory ITP patients after hUC-MSCs infusion at 7 time points, including one day before hUC-MSCs infusion, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16weeks and 28 weeks after hUC-MSCs infusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years old, male or female;
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP);
* Three months after splenectomy;
* The first-line treatment drugs such as human immunoglobulin, glucocorticoid, and the second-line treatment of thrombopoietin drugs and rituximab were invalid, or there was no response or recurrence after splenectomy;
* Diagnosis of ITP>6 months；
* More than 3 months after rituximab treatment；
* Platelet counts <30 ×10^9/L, and bleeding tendency;
* People who are willing to sign the informed consent voluntarily and follow the research program.
* Subject is practicing an acceptable method of contraception. Women of childbearing potential must have a negative serum pregnancy test in the whole study;

Exclusion Criteria:

* ECOG score standard >2；
* Secondary thrombocytopenic purpura;
* Patients with poor compliance;
* Positive serology for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), and/or hepatitis D virus (HDV), Syphilis; Positive for Epstein-Barr Virus DNA, Cytomegalovirus DNA;
* Pregnancy or lactation period;
* History of thrombosis;
* The serum chemistry results exceed the upper laboratory normal range by more than 20%, such as ALT, AST, TBIL, BUN, Cre etc;
* Pre-existing cardiac disease, including congestive heart failure of New York Heart Association [NYHA] Grade III/IV, arrhythmia requiring treatment or myocardial infarction within the last 6 months. No arrhythmia known to increase the risk of thrombotic events (e.g. atrial fibrillation), or patients with a QT >450msec or QTc > 480 for patients with a Bundle Branch Block;
* History of solid organ or bone marrow transplant;
* Researchers believe that patients should not participate in the test of any other condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of the platelet counts after hUC-MSCs infusion | 28 weeks
  The investigator will assess the changes of the platelet counts after hUC-MSCs infusion from week 1 to week 28.
Incidence of adverse events after hUC-MSCs infusion | 4 weeks
  The investigator will observe incidence of adverse events during and after hUC-MSCs infusion, including fever, thrombosis, diarrhea, skin rash and so on.
Changes in virus safety indicators after hUC-MSCs infusion | 16 weeks
  The investigator will complete virus detection( including HBV, HCV, HIV, Syphilis, EB, CMV, etc) at week 4 and week 16 after hUC-MSCs infusion.

SECONDARY OUTCOMES:
Changes of concentration of hUC-MSCs in peripheral blood | 96 hours
  The investigator will observe the concentration of hUC-MSCs in peripheral blood from female patients after the first hUC-MSCs infusion at 10 time points, including 30 minutes before hUC-MSCs infusion, 30 minutes, 60 minutes, 2 hours, 4 hours, 8 hours, 16 hours, 24 hours,48 hours and 96 hours after the first hUC-MSCs infusion.
Changes of antibody production of hUC-MSCs in peripheral blood | 24 days
  The investigator will detect antibody production of hUC-MSCs in peripheral blood from the first 9 patients at 2 time points, including 30 minutes before the first hUC-MSCs infusion and 48 hours after the last hUC-MSCs infusion.
Changes of immune function in refractory ITP patients after hUC-MSCs infusion | 28 weeks
  The investigator will observe the changes of immune function in refractory ITP patients after hUC-MSCs infusion at 7 time points, including one day before the first hUC-MSCs infusion, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16weeks and 28 weeks after the first hUC-MSCs infusion. The changes of immune function will include the changes of the percentage of Th cell subsets， regulatory T cells (Treg)，supressor T cells（Ts）, activation and proliferation of B and T lymphocyte, apoptosis of platelets by cytotoxic T cells(CTLs) and function of dendritic cells in peripheral blood mononuclear cells（PBMCs）at the 7 time points, and to compare with the healthy controls. The investigator also will assess the changes of cytokines in the cell culture supernatants and plasma at the 7 time points, and to compare with the healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Yunfei Chen, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.

REFERENCES:
- [Background] Wang X, Yin X, Sun W, Bai J, Shen Y, Ao Q, Gu Y, Liu Y. Intravenous infusion umbilical cord-derived mesenchymal stem cell in primary immune thrombocytopenia: A two-year follow-up. Exp Ther Med. 2017 May;13(5):2255-2258. doi: 10.3892/etm.2017.4229. Epub 2017 Mar 14. PMID 28565834
- [Background] Wang Y, Han ZB, Ma J, Zuo C, Geng J, Gong W, Sun Y, Li H, Wang B, Zhang L, He Y, Han ZC. A toxicity study of multiple-administration human umbilical cord mesenchymal stem cells in cynomolgus monkeys. Stem Cells Dev. 2012 Jun 10;21(9):1401-8. doi: 10.1089/scd.2011.0441. Epub 2011 Nov 22. PMID 21958114
- [Background] Wang Y, Zhang Z, Chi Y, Zhang Q, Xu F, Yang Z, Meng L, Yang S, Yan S, Mao A, Zhang J, Yang Y, Wang S, Cui J, Liang L, Ji Y, Han ZB, Fang X, Han ZC. Long-term cultured mesenchymal stem cells frequently develop genomic mutations but do not undergo malignant transformation. Cell Death Dis. 2013 Dec 5;4(12):e950. doi: 10.1038/cddis.2013.480. PMID 24309937
- [Background] Gong W, Han Z, Zhao H, Wang Y, Wang J, Zhong J, Wang B, Wang S, Wang Y, Sun L, Han Z. Banking human umbilical cord-derived mesenchymal stromal cells for clinical use. Cell Transplant. 2012;21(1):207-16. doi: 10.3727/096368911X586756. Epub 2011 Sep 16. PMID 21929848
- [Background] Wu Y, Wang Z, Cao Y, Xu L, Li X, Liu P, Yan P, Liu Z, Zhao D, Wang J, Wu X, Gao C, Da W, Han Z. Cotransplantation of haploidentical hematopoietic and umbilical cord mesenchymal stem cells with a myeloablative regimen for refractory/relapsed hematologic malignancy. Ann Hematol. 2013 Dec;92(12):1675-84. doi: 10.1007/s00277-013-1831-0. Epub 2013 Jul 11. PMID 23842707
- [Background] Liang J, Zhang H, Hua B, Wang H, Wang J, Han Z, Sun L. Allogeneic mesenchymal stem cells transplantation in treatment of multiple sclerosis. Mult Scler. 2009 May;15(5):644-6. doi: 10.1177/1352458509104590. PMID 19389752
- [Background] Wu Y, Cao Y, Li X, Xu L, Wang Z, Liu P, Yan P, Liu Z, Wang J, Jiang S, Wu X, Gao C, Da W, Han Z. Cotransplantation of haploidentical hematopoietic and umbilical cord mesenchymal stem cells for severe aplastic anemia: successful engraftment and mild GVHD. Stem Cell Res. 2014 Jan;12(1):132-8. doi: 10.1016/j.scr.2013.10.001. Epub 2013 Oct 10. PMID 24185180
- [Result] Ma L, Zhou Z, Zhang D, Yang S, Wang J, Xue F, Yang Y, Yang R. Immunosuppressive function of mesenchymal stem cells from human umbilical cord matrix in immune thrombocytopenia patients. Thromb Haemost. 2012 May;107(5):937-50. doi: 10.1160/TH11-08-0596. Epub 2012 Mar 8. PMID 22398715
- [Derived] Chen Y, Xu Y, Chi Y, Sun T, Gao Y, Dou X, Han Z, Xue F, Li H, Liu W, Liu X, Dong H, Fu R, Ju M, Dai X, Wang W, Ma Y, Song Z, Gu J, Gong W, Yang R, Zhang L. Efficacy and safety of human umbilical cord-derived mesenchymal stem cells in the treatment of refractory immune thrombocytopenia: a prospective, single arm, phase I trial. Signal Transduct Target Ther. 2024 Apr 23;9(1):102. doi: 10.1038/s41392-024-01793-5. PMID 38653983